CLINICAL TRIAL: NCT04067180
Title: Randomized Clinical Study of Haplo-Identical Donors Versus Unrelated Donors in Hematopoietic Stem Cell Transplant Patients With Acute Myeloid Leukemia
Brief Title: Randomized Clinical Study Assessing Haplo vs. URD in AML
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Delayed enrollment due to COVID-19 pandemic and other non-alterable world events, including war. The time elapsed when the study was paused has lowered the relevance of the study.
Sponsor: Karolinska Institutet (Other)
Collaborators: Skane University Hospital (Other); Uppsala University Hospital (Other); University Hospital, Linkoeping (Other); University Hospital, Umeå (Other); Sahlgrenska University Hospital (Other); Oslo University Hospital (Other); St. Petersburg State Pavlov Medical University (Other); Princess Margaret Hospital, Canada (Other); Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Jonas Mattsson, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DNR: 2017/8
Record Dates: First submitted 2019-08-20; First posted 2019-08-26 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Acute Myeloid Leukemia
Keywords: allogeneic stem cell transplantation; Haplo-identical donors; Matched unrelated donors; Alternative stem cell donors; Post-transplantation cyclophosphamide; Haplo-identical stem cell transplantation
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Haplo SCT (Experimental): Allogeneic stem cell transplantation with a haplo-identical family donor graft.
  Interventions: Other: allogeneic stem cell transplantation with a haplo-identical family donor graft
- URD SCT (Active Comparator): Allogeneic stem cell transplantation with a matched unrelated donor graft.
  Interventions: Other: allogeneic stem cell transplantation with a matched unrelated donor graft

INTERVENTIONS:
Other: allogeneic stem cell transplantation with a haplo-identical family donor graft — The graft should preferably be bone marrow, but peripheral stem cells are also acceptable.
  Pre-conditioning: thiotepa 5 mg/kg/day for two days (day -6, -5), busulfan at 3,2 mg/kg/day (i.v.) and fludarabine at 50 mg/m2 (i.v.) for three consecutive days (day -4, -3, -2). Intravenous busulfan can be replaced by orally administered busulfan at a dose of 4 mg/kg/day on 3 consecutive days (day -4, -3, -2).
  GVHD prophylaxis: cyclophosphamide 50 mg/kg day +3 and +5, cyclosporin A and mycophenolate mofetil.
  Arms: Haplo SCT
Other: allogeneic stem cell transplantation with a matched unrelated donor graft — Patients are treated according to the standard conditioning protocols developed for URD SCT at each participating center, with a recommendation to use "Flu+Bu" (fludarabine + busulfan, with a total Bu dose of 8-16 mg/kg body weight orally, or 6,4-12,8 mg/kg i.v.) or "Bu+Cy" (busulfan + cyclophosphamide, with a dose of Cy not exceeding 50 mg/kg x 2).
  The standard GVHD prophylaxis at the center should be applied.
  Arms: URD SCT

SUMMARY:
This study compares haplo-identical family donor stem cell transplantation (haplo SCT) to matched unrelated donor transplantation (URD SCT) in adult patients with acute myeloid leukemia (AML) with the hypothesis that haplo SCT is as good as URD SCT.

Background:

A haplo-identical family donor is a relative sharing 50% of the human leukocyte antigens (HLA) of the patient. SCT with this type of donor is increasing, and a number of retrospective studies have demonstrated its feasibility, but prospective randomized studies are still lacking. Such studies are necessary to establish the benefits of haplo SCT. For the ≈70% of the patients that lack the 1st choice donor, an HLA-matched sibling, the 2nd choice is an URD at most centers. However, if haplo-identical donors are as good as URDs, this could change. Haplo-identical donors have several advantages. Almost all patients have at least one available haplo-identical donor, while URDs can be difficult to find. It also eliminates the need for time-consuming donor searches, and is considerably less costly.

The Study:

Patients can be included in the study if they have AML and require SCT, ≥18 years, DO NOT have an HLA-matched sibling donor, and DO have potential haplo-identical family donors AND URDs.

After enrollment in the study, the patients are assigned randomly to either haplo SCT or URD SCT. The treatment surrounding the transplantation differs according to the donor type. Patients receiving haplo-identical transplantation are treated with a specified chemotherapy protocol before transplantation and a chemotherapy combined with immunosuppressive drugs after the transplantation to prevent graft-vs. host disease (GVHD). The patients receiving URD SCT will be treated according to the standard protocol at their center. Thus, haplo SCT will be compared to what is currently used in patients without an HLA-identical sibling today.

The primary endpoint of this study is graft-vs.-host disease- and relapse free survival two years after study inclusion. This measurement takes into account the side effect that causes the most long-term suffering, graft-vs-host disease, as well as leukemia relapse and thus indicates to what extent the treated patients remain relapse-free and without significant side effects. Secondary end points include relapse-free survival, frequencies of graft-versus-host disease and of infections, and the patients will be followed in the study for five years.

DETAILED DESCRIPTION:
This is a randomized, intention-to-treat, open label, non-inferiority study performed in an international multicenter setting comparing allogeneic stem cell transplantation (SCT) with haplo-identical family donors (haplo SCT) to matched unrelated donor (URD) SCT in adult patients with de novo or treatment related acute myeloid leukemia (AML). The primary study objective is to compare GVHD and relapse free survival (GRFS) at 2 years post-randomization in patients randomized to Haplo-SCT with patients randomized to URD-SCT.

The choice of hematopoietic stem cell donor, the humal leukocyte antigen (HLA) match, and the type of graft used are factors of major importance for survival and the risk of complications after SCT. The use of haplo-identical donors has shown very promising results and may result in a paradigm shift in SCT. However, no prospective randomized studies comparing unrelated donors, the standard choice today when no HLA-identical sibling is available, with haplo-identical donors have been published. The purpose of this study is to evaluate in a prospective and randomised fashion whether haplo-identical donor SCT could yield similar results to SCT with unrelated donors in patients with AML.

HYPOTHESIS:

The graft-vs.-host disease- and relapse-free survival two years after randomization (2-year GRFS) after haplo SCT is not inferior to 2-year GRFS after URD SCT with donors matched at 7/8 or 8/8 of the major HLA loci.

STUDY POPULATION

Adult patients with de novo or treatment-related acute myeloid leukemia with indication for allogeneic stem cell transplantation (SCT). MDS-AML and significant extramedullary AML disease is excluded to make the study population more homogeneous.

Main inclusion criteria: Adult patients (age ≥ 18 years) with de novo or treatment-related AML, eligible and fit for SCT, with at least one potential haplo-identical related donor and at least five potential HLA-A, -B, and -DRB1 antigen matched unrelated donors (URD) identified prior to inclusion.

Main exclusion criteria: Patients with a suitable HLA-identical sibling donor, and patients with less than five potential URDs, and/or without a potential haplo-identical related donor.

Sample size: The total target enrollment is 200 patients, 100 patients in each treatment arm.

STUDY PLAN

Randomization is performed when it has been determined that all inclusion criteria are fulfilled and no exclusion criteria are met. Patients will be randomized at a ratio 1:1 between the treatment arms using the permuted block technique, stratified by center to reduce geographic and recruitment location related bias.

CHOICE OF DONOR AND STEM CELL SOURCE Donors for Haplo-SCT are required to be healthy and 18-60 years of age. Siblings, children and parents are acceptable. The choice of donor is based on the clinical experience and current standard procedure at each center, taking factors such as ABO-match, presence of relevant HLA-antibodies in the recipient, cytomegalovirus (CMV)-serology compatibility, female donor to male recipient, and donor age into consideration. The presence of significant levels of HLA-antibodies against mismatched HLA molecules of the donor renders that donor unsuitable for transplantation. The primary stem cell source for Haplo-SCT in the study is bone marrow. The target dose is > 4 ×10(8) total nucleated cells (TNC)/kg patient weight. Peripheral blood stem cell grafts can be used without breaking study protocol, but is strongly discouraged in patients where bone marrow harvest of the donor is possible. If PBSC is used for Haplo-SCT in this trial, the maximum cell dose recommended is 5 ×10(6) CD34+ cells/kg patient weight.

The choice of URD is to be based on the standard donor selection algorithm and guidelines at each participating center. The chosen URD need to be allele-matched for HLA-A, -B, and -DRB1. For HLA-C, one allele or antigen mismatch is allowed. If the HLA-match between the recipient and several URDs are acceptable, other donor SCT-factors (e.g. CMV-status, ABO-compatibility, sex-match, previous pregnancies, age, weight, etc.) should be taken into consideration before the final donor choice. The choice of stem cell source (BM or PBSC) and CD34+ cell dose and total nucleated cell dose should be according to current institutional practice.

For patients randomized to either treatment arm where no suitable donor can be identified, cross over to the other arm is permitted.

TREATMENT PLAN

CONDITIONING:

Patients randomized to haplo SCT will be treated according to the Genoa protocol. This protocol is based on the administration of thiotepa 5 mg/kg/day for two days (day -6, -5), busulfan at 3,2 mg/kg/day (i.v.) and fludarabine at 50 mg/m2 (i.v.) for three consecutive days (day -4, -3, -2). Intravenous busulfan can be replaced by orally administered busulfan at a dose of 4 mg/kg/day on 3 consecutive days (day -4, -3, -2). For elderly patients (> 60 years), or patients in poor clinical condition, the dose of busulfan may be reduced (e.g. by reducing the number of treatment days, usually to 2 days for patients > 60 years old). GVHD prophylaxis for Haplo-SCT is cyclophosphamide 50 mg/kg day +3 and +5, cyclosporin A (CyA) and mycophenolate mofetil (MMF).

Patients randomized to URD SCT are treated according to the conditioning protocols used in standard practice, with a recommendation to use the conditioning regimens "Flu+Bu" (fludarabine + busulfan, with a total dose of Bu of 8-16 mg/kg body weight orally, or 6,4-12,8 mg/kg i.v.) or "Bu+Cy" (busulfan + cyclophosphamide, with a dose of Cy not exceeding 50 mg/kg x 2). If possible, all participating centers are recommended to use one myeloablative conditioning (MAC) protocol and one reduced intensity (RIC) protocol for included URD-SCT study patients throughout the study. In the majority of the participating centers, protocols including anti-thymocyte globulin (ATG) is administered. The choice of GVHD prophylaxis for the URD-SCT arm is to be performed according to the same principle as the conditioning regimen, i. e. the standard practice at the center should be applied.

IMMUNOSUPPRESSION:

The dose of CyA should be targeted and adjusted to a set serum concentration as per center preference. As a general guide, patients that have undergone Haplo-SCT could be kept at a slightly lower concentration compared to patients that have undergone URD-SCT. The guiding dosage principle is that CyA is given i.v. or p.o. at full dose from day 0 in the Haplo-SCT arm (from day -1 in the URD-SCT patients receiving CyA) to day +90 approximately, then to be tapered in the absence of GvHD and discontinued at 5-6 months after SCT or earlier if clinically indicated. Tacrolimus may replace CyA if the patient does not tolerate CyA.

In haplo SCT patients, MMF is given at 15 mg/kg x 2 orally, starting at day +1 post SCT. It is recommended to use MMF orally, but i.v. MMF is accepted. Dose adjustment is necessary in patients suffering from severely impaired kidney or liver function. MMF is discontinued day +28. In case MMF is used in URD-SCT patients, this is to be done according to the standard protocols of the transplant center concerned.

Other relevant GVHD prophylaxis strategies for URD-SCT are also permitted.

SUPPORTIVE CARE

Supportive care is to be performed according to standard procedure at each participating center.

FOLLOW UP

Patients will be followed for GRFS, survival, relapse, and other listed end-points at designated time points. The primary endpoint will be reached when the last included patient has a follow-up time of 2 years. The study will be terminated when the last included patient has a follow-up time of five years. Data collection is continued even if the assigned therapy was not carried out, since the main study analyses are intention-to-treat analyses. Per-protocol analyses will be performed as well.

STUDY-SPECIFIC SAMPLES

Study samples from peripheral blood:

Study samples from peripheral blood are requested at the visit for randomization, at the day of SCT-graft infusion (day 0), and at follow-up visits after 1, 3, 6, 12 and 24 months post-SCT. At all of these time-points,

Study samples from bone marrow:

Study samples from bone marrow aspiration material are requested at the follow-up visits after 2-3, 6, 12 and 24 months post-SCT (see Appendix IV for reference). At all of these time-points,

STUDY MANAGEMENT

Source data and data management Data will be collected continuously and entered into the study specific electronic case report form (eCRF). Study-related documents will be retained for at least 25 years.

Quality control and monitoring The study will be monitored regularly according to good clinical practice (GCP) and local regulations to ensure accurate, complete and reliable data. All information reported in the eCRF will also be documented in the patient's file unless otherwise specified.

Patient information and consent Before inclusion patients will receive verbal and written information including a description of the trial, its purpose, the risks and the procedures involved. Written informed consent must be obtained from all patients before enrollment in the study.

Adverse Event (AE) Reporting Reported in the eCRF according to CTCAE version 4.03.

Serious Adverse Event (SAE) reporting For the purpose of this study, SAEs that are regarded as expected events considering the given treatment (i.e. allogeneic hematopoietic stem cell transplantation) and underlying disease, need not be reported as SAEs. However, all deaths and unexpected significant SAEs are to be reported.

Study Safety Board A Study Safety Board (SSB) will perform safety analyses during the study. This is a study independent data-monitoring committee that is established by the Sponsor to assess at intervals the progress of the clinical trial, the safety data, and the critical endpoints of the trial. The SSB will consist of three members, with at least one independent statistician and two internationally renowned clinical hematologists.

The SSB will receive at least the following reports from the trial statistician for review:

* Interim analysis reports when 50% of the patients have been included, and when 100% of the patients have been included in the trial.
* Annual safety data listing the incidence of (serious) adverse events.
* Annual progress data listing the number of enrolled patients and the status of data collection.

Study termination and stopping rules

Regular study termination The study will be terminated when the last included surviving patient has a follow-up of five years in the trial.

Stopping rules Termination of the study will be considered if, at the first interim analysis, the rate of non-relapse mortality (NRM) ≥ 40% at 200 days after SCT, and/or the rate of acute GVHD grades III-IV ≥ 20% in evaluable patients (with sufficient follow-up time or evaluation) in the Haplo-SCT arm.

ELIGIBILITY:
Inclusion Criteria:

* 1. Adult patients (age ≥ 18 years) with de novo or treatment-related AML, eligible and fit for SCT treatment according to national/international guidelines.
* 2. One or more potential haplo-identical related donor(s) AND five or more potential 6/6 HLA-A, -B, and -DRB1 antigen matched unrelated donors identified before randomization.
* 3. Karnofsky Performance Status ≥ 70% at randomization.
* 4. Signed informed consent.
* 5. Patient willing and able to comply with protocol requirements

Exclusion Criteria:

* 1. Patients with a suitable HLA-identical sibling donor.
* 2. Patients with < 5 potential HLA-A, -B, and -DRB1 antigen matched URDs available.
* 3. Patients with no potential haplo-identical related donor available.
* 4. Patients scheduled for/receiving cord blood stem cell transplantation.
* 5. Prior allogeneic SCT using any hematopoietic stem cell source.
* 6. Patients seropositive for HIV.
* 7. Pregnancy (positive β-HCG test) within 4 weeks of study entry.
* 8. Cardiac ejection fraction < 45%.
* 9. Karnofsky Performance Status < 70% at time of randomization.
* 10. The presence of any psychological, family-related, social, and/or geographical condition potentially jeopardizing compliance with the study protocol and follow-up schedule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2022-08-26 (Actual); Study Completion 2022-08-26 (Actual)

PRIMARY OUTCOMES:
Intention to treat analysis of 2-year graft-vs.-host disease- and relapse-free survival | 2 years
  Defined in this study as the time between inclusion and either grades III-IV acute GVHD, severe chronic GVHD or disease relapse. All events occuring from SCT to last follow-up are considered when calculating GRFS. Incomplete data resulting from patients who are lost to follow-up or who withdraw their informed consent will be censored at the date they were last known to be alive. Patients who are alive at study termination will be censored at the latest date of contact. Analysed according to original treatment arm assignment (intention-to-treat)

SECONDARY OUTCOMES:
Per protocol analysis of 2-year graft-vs.-host disease- and relapse-free survival | 2 years
  The time between inclusion and either grades III-IV acute GVHD, severe chronic GVHD or disease relapse. Analysed according to received treatment (per protocol)
Intention to treat analysis of 5-year graft-vs.-host disease- and relapse-free survival | 5 years
  The time between inclusion and either grades III-IV acute GVHD, severe chronic GVHD or disease relapse. Intention to treat analysis.
Per protocol analysis of 5-year graft-vs.-host disease- and relapse-free survival | 5 years
  The time between inclusion and either grades III-IV acute GVHD, severe chronic GVHD or disease relapse. Per protocol analysis.
Intention to treat analysis of Overall survival | 2 years and 5 years
  Defined as the time interval between the date of study inclusion and the date of death from any cause. Incomplete data resulting from patients who are lost to follow-up or who withdraw their informed consent will be censored at the date they were last known to be alive. Patients who are alive at study termination will be censored at the latest date of contact. Analysed according to original treatment arm assignment (intention-to-treat)
Intention to treat analysis of Disease-free survival | 2 years and 5 years
  The time between date of inclusion and date of relapse or death from any cause. Incomplete data resulting from patients who are lost to follow-up or who withdraw their informed consent will be censored at the date they were last known to be alive. Patients who are alive at study termination will be censored at the latest date of contact. Analysed according to original treatment arm assignment (intention-to-treat)
Per protocol analysis of Overall survival | 2 years and 5 years
  Defined as the time interval between the date of study inclusion and the date of death from any cause. Analysed according to received treatment (per protocol)
Per protocol analysis of Disease-free survival | 2 years and 5 years
  Defined as the time between date of inclusion and date of relapse or death from any cause.. Analysed according to received treatment (per protocol)
Acute graft.vs.-host disease | 2 years
  Cumulative incidence of acute graft-vs.-host disease grades I-IV
Chronic graft.vs.-host disease | 2 years and 5 years
  Cumulative incidence of chronic graft-vs.-host disease
Infection | 2 years
  Cumulative incidence of infectious complications after transplantation, including bacterial blood-stream infections, fungal infections, viral infections such as cytomegalovirus and Epstein-Barr virus and other infections.
Relapse | 2 years and 5 years
  Relapse of the patients
Engraftment of neutrophil granulocytes | 90 days
  Cumulative incidence of neutrophil granulocyte engraftment (defined as reaching ≥0.5 x 10(9)/L in peripheral blood) after transplantation.
Engraftment of thrombocytes | 1 year
  Cumulative incidence of thrombocyte engraftment (defined as reaching ≥30 and ≥50 x 10(9)/L in peripheral blood) after transplantation.
Other non-specified transplant complications | 2 years
  A wide variety of transplant complications are known to occur, such as organ damage and organ failure due to the conditioning and other transplant-related treatments. The occurrence of such will be analysed.
Secondary malignancies | 5 years
  The development of malignancies after transplantation, excluding relapse of the original AML the patient received transplantation for.

CONTACTS AND LOCATIONS:
Overall Officials: Johan Karlsson Torlen, MD PhD, Study Chair — Karolinska Institutet
Locations (9):
- Medical University of Vienna, Vienna, Austria
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada
- Oslo University Hospital, Oslo, Norway
- Pavlov First Saint-Petersburg State Medical University, Saint Petersburg, Russia
- Sweden (5):
  - Sahlgrenska University Hospital, Gothenburg
  - Linköping University Hospital, Linköping
  - Skåne University Hospital, Lund
  - Umeå University Hospital, Umeå
  - Uppsala University Hospital, Uppsala